CLINICAL TRIAL: NCT05707715
Title: Comfort and Support Values Provided by Different Pillow Designs for Individuals With Forward Head Posture
Brief Title: Comfort and Support Values of Different Pillow Designs
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Ceyhun Türkmen, Asst. Prof., Çankırı Karatekin University
Other Study IDs: 19/01/2023-30
Record Dates: First submitted 2023-01-22; First posted 2023-02-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Sleep; Proprioceptive Disorders; Orthopedic Disorder
MeSH Terms: conditions — Somatosensory Disorders; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Slight Forward Head Posture: This descriptive cross-sectional study which was approved by Çankırı Karatekin University Ethics Committee (Approval number:). There is FHP if the imaginary line between the tragus of the ear and the middle of the shoulder is not on the same line when viewed from the side. And the horizontal length between that two vertical lines indicates the severity of FHP. The level of FHP is classified as slight/severe/highly FHP according to that horizontal length. The slight FHP is accepted as between 0-2.5cm, and severe FHP above 2.5cm (27).
  Interventions: Device: XSensor
- Severe Forward Head Posture: This descriptive cross-sectional study which was approved by Çankırı Karatekin University Ethics Committee (Approval number:). There is FHP if the imaginary line between the tragus of the ear and the middle of the shoulder is not on the same line when viewed from the side. And the horizontal length between that two vertical lines indicates the severity of FHP. The level of FHP is classified as slight/severe/highly FHP according to that horizontal length. The slight FHP is accepted as between 0-2.5cm, and severe FHP above 2.5cm (27).
  Interventions: Device: XSensor

INTERVENTIONS:
Device: XSensor — A pressure mapping system (X3 SENSOR PX 100:64.160.02, X-Sensor®, Calgary, Canada) was used to record the pressure distribution in mmHg of the head and shoulder section [18,19]. Pressure distribution was recorded for 1 minute for each lying position. The purpose of these measurements was to describe the pressure distribution created by the participants in the pillow and the supported areas, as well as to find out the differences that may occur between the pillows. Lower pressure values measured by the device were defined as "high comfort", while more contact of the head area with the pillow was accepted as "high support".

SUMMARY:
With the change in lifestyle, most physical tasks are now performed by machines. As a result, sitting has become the most common learning posture and office posture, and cervical and lumbar spondylosis are becoming increasingly prevalent in younger people. One-third of life is devoted to sleep, and bad sleeping posture can place incorrect strain on the cervical and lumbar spine, resulting in irreversible and detrimental repercussions if not treated seriously. Sleep disorders have become an important public health concern because they can have detrimental effects on both mental and physical health. A pillow can give adequate support for the head and neck and assist sleepers in maintaining proper neck and thoracic curvature. Studies have demonstrated that a comfortable sleeping pillow helps relax the neck muscles, hence facilitating sleep, and efficiently alleviate pain in the neck, shoulders, back, and head.

There is consensus among researchers that supporting the natural lordotic curve of the cervical spine is necessary to achieve longer periods of deep sleep. In addition, a pillow can improve sleep quality by cooling the head, lowering body temperature, reducing sweating or slowing the heart rate during sleep. However, the level of evidence to support these claims is so far limited. It has been claimed by pillow manufacturers that many design-related pillow parameters are effective in improving sleep quality and reducing neck pain. However, most of these recommendations are based on personal experience.

This study recommends the most suitable pillow for people in forward head postures based on the body pressure distribution of the head, neck and upper body. The proposed pillows were evaluated in two parameters: comfort and support.

DETAILED DESCRIPTION:
With the change in lifestyle, most physical tasks are now performed by machines. As a result, sitting has become the most common learning posture and office posture, and cervical and lumbar spondylosis are becoming increasingly prevalent in younger people. One-third of life is devoted to sleep, and bad sleeping posture can place incorrect strain on the cervical and lumbar spine, resulting in irreversible and detrimental repercussions if not treated seriously. Sleep disorders have become an important public health concern because they can have detrimental effects on both mental and physical health. A pillow can give adequate support for the head and neck and assist sleepers in maintaining proper neck and thoracic curvature. Studies have demonstrated that a comfortable sleeping pillow helps relax the neck muscles, hence facilitating sleep, and efficiently alleviate pain in the neck, shoulders, back, and head.

While studies on the support and comfort of human contact surfaces generally focus on sitting posture, there is limited information available because the assessment of sleep position is more complex. The main reason behind this confusion is that the human body can take many different positions while sleeping. In supine, prone or side lying positions, the pressure or support properties of the human contact surfaces of the pillow against individuals vary greatly. In addition, head-neck curvatures that vary from person to person can also change their support and comfort needs.

In current research on pillows, assessments can be made subjectively or objectively. Subjective evaluations are made by completing an evaluation form based on the person's self-report after the sleep test. In this evaluation form, the amount of comfort and support that the person gets from the pillow is questioned. Although this method directly reveals one's own thoughts, it has poor reproducibility, the results can be easily manipulated, it takes a long time to be done, and it is not suitable for complex experiments. Objective assessments can be made by analyzing body pressure distributions, EMG signals and anthropometric characteristics of individuals. According to the results of the studies, it has been shown that the evaluation method performed with body pressure distributions is the most effective method. This may be because body pressure distribution can respond quickly to materials used, support arrangements, human weight or lying positions.

Studies have shown that long-term high pressure applied to certain parts of the human body can affect the human central nervous, blood circulatory and endocrine system. In addition, different parts of the human body show great sensitivity to pressure due to differences in subcutaneous tissue and tissue structures. In terms of ergonomics, the pressure perception of the human body can be divided into dull parts and sensitive parts. Dull parts can withstand more pressure, while sensitive parts can only feel comfortable when the pressure is low. Therefore, one of the main goals in pillow selection should be to reduce the pressure applied to sensitive points.

Although it has been reported that the main role of the pillow is to optimize head and neck posture, there are limited studies on its effectiveness in terms of its effect on head and neck posture. About a third of human life is spent in sleep, during which the spine is beyond our conscious control. Therefore, pillows play an important role in maintaining ideal head and neck posture and can change muscle activities.

Head and neck position is an important factor affecting sleep quality. It is reported that while sleeping, cervical control weakens and places excessive stress on spinal structures. Symptoms such as neck and shoulder pain, tension headaches and muscle stiffness that occur during this time reduce sleep quality. That's way, there is a serious requirement to investigate how different pillow designs can effectively support the cervical spine to reduce neck pain and thus improve sleep quality.

Forward head posture (FHP) is the anterior alignment of the cervical spine; it is also known as "text neck," "scholar's neck," "wearies neck," "ihunch," and "reading neck." Several factors, including sleeping with the head lifted excessively high, prolonged use of computers, laptops, and cell phones, lack of developed back muscle strength, and nutritional deficiencies such as calcium, contribute to this postural disorder. Age is linked with decreased cervical ROM, thoracic kyphosis is associated with increased cervical flexion, and increased forward head posture is associated with larger deficits in cervical rotation and flexion ROM.

Scientific evidence suggests that head postural changes affect the development and persistence of neck pain. Therefore, it should be one of the main factors for choosing an ergonomically correct pillow. In addition, the cervical muscles play an important role in the control of neck posture. The reduced ability of these muscles to maintain the upright posture of the cervical spine may indicate that their endurance is impaired and they are unable to maintain cervical lordosis. Since various studies often report a significant association between weak neck muscles, poor posture, and experience of neck pain, and considering that a pillow can reduce pain and disability, it should be considered that the pillow needs of individuals with a forward head posture may differ.

Pillow comfort research is relatively new and the factors affecting the selection of the right pillow are still unclear. For example, it is not correct to accept the head and neck regions as a whole and accept comfort and support demands as similar. Because the position of the head with respect to the height differs in the normal head posture or tilting the head forward, and this may affect the comfort or support properties of the pillow. Due to differences in head posture, the comfort and support demands of the head and neck areas in contact with the pillow will also vary.

There is consensus among researchers that supporting the natural lordotic curve of the cervical spine is necessary to achieve longer periods of deep sleep. In addition, a pillow can improve sleep quality by cooling the head, lowering body temperature, reducing sweating or slowing the heart rate during sleep. However, the level of evidence to support these claims is so far limited. It has been claimed by pillow manufacturers that many design-related pillow parameters are effective in improving sleep quality and reducing neck pain. However, most of these recommendations are based on personal experience.

This study recommends the most suitable pillow for people in forward head postures based on the body pressure distribution of the head, neck and upper body. The proposed pillows were evaluated in two parameters: comfort and support.

ELIGIBILITY:
Inclusion Criteria:

* Forward head posture
* Good cognitive status (Mini Mental Test >23/30

Exclusion Criteria:

* Orthopeadical or Neurological chronic disorders
* Spinal disraphism
* Spinal rheumotological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-22 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Comfort and support assessment | 15 minutes
  A pressure mapping system (X3 SENSOR PX 100:64.160.02, X-Sensor®, Calgary, Canada) was used to record the pressure distribution in mmHg of the head and shoulder section [18,19]. The pressure mapping system used has a sensing area of 81.3 × 203.2 cm (32'' x 80''), provides high resolution sensing (1.27 cm or 0.5'') using 10,240 sensing points with an accuracy of ±2 mmHg. For the purpose of our study, the pressure mapping system was positioned on the pillow and the patients were asked to lie on the mapping system once in supine, side lying and prone positions. The purpose of these measurements was to describe the pressure distribution created by the participants in the pillow and the supported areas, as well as to find out the differences that may occur between the pillows. Lower pressure values measured by the device were defined as "high comfort", while more contact of the head area with the pillow was accepted as "high support".

CONTACTS AND LOCATIONS:
Locations (1):
- ODTU Teknopark ASO, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andreoni G, Santambrogio GC, Rabuffetti M, Pedotti A. Method for the analysis of posture and interface pressure of car drivers. Appl Ergon. 2002 Nov;33(6):511-22. doi: 10.1016/s0003-6870(02)00069-8. PMID 12507335
- [Result] Le P, Rose J, Knapik G, Marras WS. Objective classification of vehicle seat discomfort. Ergonomics. 2014;57(4):536-44. doi: 10.1080/00140139.2014.887787. Epub 2014 Mar 7. PMID 24606493
- [Result] de Looze MP, Kuijt-Evers LF, van Dieen J. Sitting comfort and discomfort and the relationships with objective measures. Ergonomics. 2003 Aug 15;46(10):985-97. doi: 10.1080/0014013031000121977. PMID 12850935
- [Result] Miyatsuji A, Matsumoto T, Mitarai S, Kotabe T, Takeshima T, Watanuki S. Effects of clothing pressure caused by different types of brassieres on autonomic nervous system activity evaluated by heart rate variability power spectral analysis. J Physiol Anthropol Appl Human Sci. 2002 Jan;21(1):67-74. doi: 10.2114/jpa.21.67. PMID 11938611
- [Result] Zhong S, Shen L, Zhou L, Guan Z. Predict human body indentation lying on a spring mattress using a neural network approach. Proc Inst Mech Eng H. 2014 Aug;228(8):787-99. doi: 10.1177/0954411914547552. Epub 2014 Aug 22. PMID 25150192
- [Result] Leilnahari K, Fatouraee N, Khodalotfi M, Sadeghein MA, Kashani YA. Spine alignment in men during lateral sleep position: experimental study and modeling. Biomed Eng Online. 2011 Nov 30;10:103. doi: 10.1186/1475-925X-10-103. PMID 22129355
- [Result] Diab AA, Moustafa IM. The efficacy of forward head correction on nerve root function and pain in cervical spondylotic radiculopathy: a randomized trial. Clin Rehabil. 2012 Apr;26(4):351-61. doi: 10.1177/0269215511419536. Epub 2011 Sep 21. PMID 21937526